CLINICAL TRIAL: NCT05005182
Title: Phase II Study to Determine the Efficacy and Safety of Luspatercept (ACE-536) in Patients With Myelodysplastic/Myeloproliferative Neoplasms With Ring Sideroblasts and Thrombocytosis (MDS/MPN-RS-T) and Myelodysplastic/Myeloproliferative Neoplasms, Unclassifiable With Ring Sideroblasts (MDS/MPN-U With RS)
Brief Title: Luspatercept With or Without Hydroxyurea for the Treatment of Myelodysplastic/Myeloproliferative Neoplasms With Ring Sideroblasts and Thrombocytosis or Unclassifiable With Ring Sideroblasts
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC200805; NCI-2021-08519 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-013021 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-08-09; First posted 2021-08-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasm With Ring Sideroblasts and Thrombocytosis, Not Otherwise Specified; Myelodysplastic/Myeloproliferative Neoplasm, Not Otherwise Specified
MeSH Terms: conditions — Thrombocytosis; Myeloproliferative Disorders | interventions — Specimen Handling; Biopsy; Hydroxyurea; luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (luspatercept) (Experimental): Patients receive luspatercept SC on day 1. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow biopsy and aspirate at baseline and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Biological: Luspatercept; Other: Questionnaire Administration
- Cohort A (luspatercept, hydroxyurea) (Experimental): Patients receive luspatercept SC on day 1 and hydroxyurea PO on days 1-21. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow biopsy and aspirate at baseline and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Hydroxyurea; Biological: Luspatercept; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspirate
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Hydroxyurea — Given PO
  Other Names: Droxia; Hydrea; Hydroxycarbamide; Litalir; Onco-Carbide; Oncocarbide; Oxeron; SQ 1089; SQ-1089; Syrea; WR 83799
  Arms: Cohort A (luspatercept, hydroxyurea)
Biological: Luspatercept — Given SC
  Other Names: ACE-536; Luspatercept-aamt; Reblozyl
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effects of luspatercept with or without hydroxyurea in treating patients with myelodysplastic/myeloproliferative neoplasms with ring sideroblasts and thrombocytosis or unclassifiable with ring sideroblasts. Biological therapies, such as luspatercept, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Hydroxyurea may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving luspatercept with or without hydroxyurea may help doctors determine what doses of the combination is safe for patients to take and how the disease responds to the treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To document the erythroid response rate assessed as per the 2015 International Working Group (IWG) myelodysplastic (MDS)/myeloproliferative neoplasms (MPN) response criteria.

SECONDARY OBJECTIVES:

I. To document response duration, time to acute myeloid leukemia (AML) transformation, AML-free survival (LFS) and overall survival (OS) in patients with MDS/MPN-with ring sideroblasts (RS) and thrombocytosis (T) and MDS/MPN-unclassifiable (U)U with RS.

II. To document safety of luspatercept (luspatercept-aamt) in patients with MDS/MPN-RS-T and MDS/MPN-U with RS.

EXPLORATORY OBJECTIVE:

I. To assess overall health-related quality of life as measured by Hematological Malignancy Specific Patient-Reported Outcome Measure (HM-PRO).

CORRELATIVE RESEARCH OBJECTIVE:

I: To find an effective biomarker of response to luspatercept-aamt.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive luspatercept subcutaneously (SC) on day 1. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow biopsy and aspirate at baseline and on study.

COHORT B: Patients receive luspatercept SC on day 1 and hydroxyurea orally (PO) on days 1-21. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow biopsy and aspirate at baseline and on study.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Patients with a World Health Organization(WHO)-defined diagnosis of MDS/MPN-RS-T or MDS/MPN-U with >= 15% RS
* Prior treatment with lenalidomide, hypomethylating agents, immunosuppressive therapy, erythropoietin stimulating agents (ESA) or investigational agent is allowed as long as patients have not received luspatercept-aamt or sotatercept. If there is prior history of investigational agent, there should be an interval equivalent to at least four elimination half-lives of the agent prior to enrollment. Note: For patients who have received prior lenalidomide, hypomethylating agents, or immunosuppressive therapy, there must be >= 6 weeks since the last dose before luspatercept-aamt treatment is started
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2
* Requirement of red blood cell transfusions (>= 2 unit =< 8-weeks prior to registration) OR symptomatic anemia with hemoglobin < 9.5 g/dL OR hematocrit < 30% (as long as there is documentation of adequate iron stores (ferritin > 50 mg/L) =< 5 weeks prior to registration). Symptomatic anemia is defined as fatigue with or without exertion, shortness of breath with or without exertion, or decrease in exercise tolerance
* Hemoglobin =< 9.5 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 30 ml/min using the Cockcroft-Gault (obtained =< 14 days prior to registration)
* Females of childbearing potential (FCBP) defined as a sexually mature woman who:

  * Has achieved menarche at some point
  * Has not undergone a hysterectomy or bilateral oophorectomy, or
  * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) and must:

    * Must have two negative urine or serum pregnancy tests as verified by the investigator prior to starting study therapy. A negative pregnancy test must be done =< 7 days prior to registration. Patient must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence from heterosexual contact
    * Either commit to true abstinence*from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with highly effective, contraception without interruption during the study therapy (including dose interruptions), and for 84 days after discontinuation of study therapy

      * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male participants must:

  * Practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 84 days following investigational product discontinuation even if he has undergone a successful vasectomy

    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willingness to provide mandatory blood specimens for correlative research

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ highly effective contraception
* Any of the following prior therapies:

  * Surgery =< 3 weeks prior to registration
  * Chemotherapy or other agents =< 2 weeks prior to registration
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Uncontrolled hypertension (defined as systolic blood pressure >= 140 mmHg or diagnostic blood pressure >= 90 mmHg despite use of >= 3 anti-hypertensive drugs at optimal doses)
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Clinically significant (symptomatic) anemia either due to nutritional deficiencies or iron, vitamin B12, folate or gastrointestinal (GI) bleeding
  * Any other conditions that would limit compliance with study requirements
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state (CD4 =< 200 x 10^6/L), are eligible for this trial
* Receiving any other drug (except hydroxyurea) or investigational agent which would be considered as a treatment for the primary disease, that is, MDS/MPN-RS-T or MDS/MPN-U with RS =< 2 weeks prior to registration
* Other active malignancy =< 3 years prior to registration. Patients on hormonal therapy for treated breast or prostate cancer are permitted if they meet other eligibility criteria

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (luteinizing hormone-releasing hormone (LHRH) agonists for prostate cancer, and treatment with bisphosphonates and receptor activator of nuclear factor kappa-B ligand [RANKL] inhibitors) for their cancer
* History of myocardial infarction, stroke, embolism, deep vein or arterial thrombosis =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek A. Mangaonkar, M.B.B.S., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Patnaik MM, Tefferi A. Luspatercept use for lower risk myelodysplastic syndromes: Active but not enough. Am J Hematol. 2023 Aug;98(8):1171-1175. doi: 10.1002/ajh.27003. Epub 2023 Jun 22. No abstract available. PMID 37345627
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Luspatercept): Patients receive luspatercept SC on day 1. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity.
- Cohort B (Luspatercept, Hydroxyurea): Patients receive luspatercept SC on day 1 and hydroxyurea PO on days 1-21. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients have been combined in order to maintain patient privacy
Groups:
- All Patients: Cohort A (luspatercept) patients receive luspatercept SC on day 1. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity.>
  > Cohort B (luspatercept, hydroxyurea) patients receive luspatercept SC on day 1 and hydroxyurea PO on days 1-21. Cycles repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Patients
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Erythroid Response Rate
Description: Defined as the proportion of patients who achieve an erythroid response out of the total number of evaluable patients (i.e. eligible patients who received at least one dose of treatment on study).
Time Frame: 8 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
Number analyzed (Participants) | 1 | 2
proportion of participants | 0 | 0.5

2. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: AEs as well as toxicities (AEs felt to be at least possibly related to study treatment) will be reported in the adverse events section of the report. The count of participants by cohort that were evaluated for address events is reported here.
Time Frame: 3 months, 29 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

3. Secondary Outcome: Duration of Response
Description: Time from erythroid response to progression or death.
Time Frame: 69 days
Population: All patients that achieved Erythroid response.
Measure: Number; unit: Days
Arm/Group | Cohort B (Luspatercept, Hydroxyurea)
Number analyzed (Participants) | 1
Days | 69

4. Secondary Outcome: Time to Leukemic Transformation
Description: Will be evaluated and characterized within each cohort using the methods of Kaplan and Meier.
Time Frame: 6 months
Population: No AML transformations were reported among the three patients on trial.
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Leukemia-free Survival
Description: Will be evaluated and characterized within each cohort using the methods of Kaplan and Meier.
Time Frame: From time of treatment to progression to acute myeloid leukemia or death from any cause, assessed up to 6 months
Population: No AML transformations were reported among the three patients on trial.
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival
Description: Will be evaluated and characterized within each cohort using the methods of Kaplan and Meier.
Time Frame: 117 117 days [was intended to be 'Up to 6 months' (duration of treatment), but study terminated early due to slow accrual]
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
Number analyzed (Participants) | 1 | 2
days | 87.0 [NA to NA] — Not enough events or patients to calculate the confidence intervals | NA [NA to NA] — Not enough events to calculate the median or confidence intervals

ADVERSE EVENTS:
Time Frame: 3 months, 29 days
Arm/Group | Cohort A (Luspatercept) | Cohort B (Luspatercept, Hydroxyurea)
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Luspatercept) (N=1) | Cohort B (Luspatercept, Hydroxyurea) (N=2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Luspatercept) (N=1) | Cohort B (Luspatercept, Hydroxyurea) (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1)
Fever (General disorders) | 1 (2) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (7) | 0 (0)
White blood cell decreased (Investigations) | 1 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decr lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT05005182/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT05005182/ICF_001.pdf